CLINICAL TRIAL: NCT05996198
Title: A Pilot Proof of Concept, Single Site Study to Assess the Effect of Exoskeletal Support on Motor Control Strategies in Individuals With Stroke
Brief Title: Exoskeletal Support in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00842
Record Dates: First submitted 2023-08-09; First posted 2023-08-18 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exoskeleton Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Patients with History of Stroke (Experimental): Individuals with history of stroke more than 6 months prior to enrollment.
  Participants will complete 3 blocks of 54 trials in a single session. Block 1 is a baseline phase where subjects will perform reaches without any loads applied via the exoskeleton devices. Block 2 is the intervention block where bilateral exoskeletons apply gravity assistance to the impaired arm for stroke survivors and gravity resistance to the non-impaired arm. Block 3 is a retention block, where tested procedures are identical to block 1.
  Interventions: Device: Oculus Rift headset; Device: Exoskeleton Device
- Healthy Controls (Experimental): Healthy age and gender-matched control participants.
  Participants will complete 3 blocks of 54 trials in a single session. Block 1 is a baseline phase where subjects will perform reaches without any loads applied via the exoskeleton devices. Block 2 is the intervention block where bilateral exoskeletons apply gravity assistance to the non-dominant arm and resistance is applied to the dominant arm in healthy controls. Block 3 is a retention block, where tested procedures are identical to block 1.
  Interventions: Device: Oculus Rift headset; Device: Exoskeleton Device

INTERVENTIONS:
Device: Oculus Rift headset — The Oculus Rift is a commercially-available virtual reality (VR) headset. It is used to present the visual environment in which participants perform the reaching task.
Device: Exoskeleton Device — The exoskeleton was designed and constructed to provide either gravity assistance or gravity resistance. It applies a torque to both shoulders. Torque values do not exceed 50% of the torque due to gravity. The device is mounted to a testing chair and attached to the participant using Velcro straps.

SUMMARY:
This interventional study will measure motor performance, including 3D movement analysis and muscle activity, in response to exoskeleton assistance. The cohort design will compare stroke patients to healthy controls. Data collection will be conducted in a single, 2-hour session. Investigators will also access stroke patients' brain MRIs that were obtained as standard of care during acute admission for stroke.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls:

* Having obtained the age of 18 years
* Neurologically healthy (i.e., no history of: traumatic brain injury, peripheral neuropathy, seizures, etc.)
* Strongly right-handed according to at least 80% score on the Edinburgh Handedness Inventory (Oldfield, 1971; Veale, 2013). The use of right-handed participants is a common feature in this field of study. This is due to the slight differences in arm control between left- and right-handed individuals (Sainburg & Kalakanis, 2000).
* Ability to give informed consent

Survivors of stroke:

* Having obtained the age of 18 years
* have a diagnosis of stroke more than six months prior to entry into the study;
* have the ability to reach, unsupported, to approximately 70% of arm length
* ability to give informed consent

Exclusion Criteria:

All participants

* have any conditions that limit their capability of using a Head Mounted Display (HMD) for a VR environment or cooperate with the protocol.
* have any orthopedic injuries to the upper extremities.
* Have neurological injuries other than stroke.
* Have excessive pain in any joint of either arm that could limit the ability to cooperate with the protocols.
* Visuospatial neglect
* Apraxia
* Global inattention
* Legal blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Schambra, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health (222 East 41st Street), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Alexander Brunfeldt, PhD [alexander.brunfeldt@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Alexander Brunfeldt, PhD [alexander.brunfeldt@nyulangone.org]. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With History of Stroke: Individuals with history of stroke more than 6 months prior to enrollment.
  Participants will complete 3 blocks of 54 trials in a single session. Block 1 is a baseline phase where subjects will perform reaches without any loads applied via the exoskeleton devices. Block 2 is the intervention block where bilateral exoskeletons apply gravity assistance to the impaired arm for stroke survivors and gravity resistance to the non-impaired arm. Block 3 is a retention block, where tested procedures are identical to block 1.
  Oculus Rift headset: The Oculus Rift is a commercially-available virtual reality (VR) headset. It is used to present the visual environment in which participants perform the reaching task.
  Exoskeleton Device: The exoskeleton was designed and constructed to provide either gravity assistance or gravity resistance. It applies a torque to both shoulders. Torque values do not exceed 50% of the torque due to gravity. The device is mounted to a testing chair and attached to the participant using Velcro straps.
- Healthy Controls: Healthy age and gender-matched control participants.
  Participants will complete 3 blocks of 54 trials in a single session. Block 1 is a baseline phase where subjects will perform reaches without any loads applied via the exoskeleton devices. Block 2 is the intervention block where bilateral exoskeletons apply gravity assistance to the non-dominant arm and resistance is applied to the dominant arm in healthy controls. Block 3 is a retention block, where tested procedures are identical to block 1.
  Oculus Rift headset: The Oculus Rift is a commercially-available virtual reality (VR) headset. It is used to present the visual environment in which participants perform the reaching task.
  Exoskeleton Device: The exoskeleton was designed and constructed to provide either gravity assistance or gravity resistance. It applies a torque to both shoulders. Torque values do not exceed 50% of the torque due to gravity. The device is mounted to a testing chair and attached to the participant using Velcro straps.
Period: Overall Study
Arm/Group | Patients With History of Stroke | Healthy Controls
Started | 9 | 10
Completed | 8 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With History of Stroke | Healthy Controls | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.75 (8.46) | 61.6 (11.49) | 60.77 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Relative Contribution (RC)
Description: Relative Contribution (RC) is a measure of the relative displacement between the hands during a bimanual reaching task. Displacement of both hands was measured using 3D motion capture using the Oculus Rift VR system. RC is calculated as the displacement of the more-impaired hand divided by the sum of displacements of both hands, multiplied by 100.
Time Frame: End of VR Task (Day 1 - session lasts approx. 2 hours)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Patients With History of Stroke | Healthy Controls
Number analyzed (Participants) | 8 | 10
percent | -0.74 (1.94) | -0.25 (1.65)

2. Primary Outcome: Muscle Contribution (MC)
Description: Muscle Contribution (MC) is a measure of the relative muscle activity between the arms during a bimanual reaching task. Muscle activity was measured using electromyography (EMG); the root-mean-square (RMS) of the EMG timeseries signal in the anterior deltoid. MC in the anterior deltoid was calculated as the RMS in the more-impaired anterior deltoid divided by the sum of RMS values in both anterior deltoids, multiplied by 100. For example, an MC (deltoid) value of 50% indicates that the muscle activity in both anterior deltoids was the same while reaching; an MC value less than 50% indicates that reaching occurred with less muscle activity in the more-impaired deltoid compared to the less-impaired deltoid.
Time Frame: Baseline, End of VR Task (Day 1 - session lasts approx. 2 hours)
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Patients With History of Stroke | Healthy Controls
Number analyzed (Participants) | 8 | 10
Percent | -0.68 (2.86) | -4.35 (11.58)

3. Secondary Outcome: Corticospinal Tract (CST) Lesion Load
Description: Measured via MRI; lesion load is expressed as percentage of the entire CST.
Time Frame: Baseline
Population: Outcome Measure was not assessed for the "Healthy Control" Arm/Group as the healthy controls do not have lesioned brain tissue.
Measure: Mean (Standard Deviation); unit: Percentage of the entire CST
Arm/Group | Patients With History of Stroke | Healthy Controls
Number analyzed (Participants) | 7 | 0
Percentage of the entire CST | 5.71 (6.6) |

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Patients With History of Stroke | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT05996198/Prot_SAP_000.pdf